CLINICAL TRIAL: NCT01283724
Title: A Multi-center, Open Label, Single-arm Study to Investigate the Safety and Efficacy of Daily Oral Administration of 2 mg Dienogest Tablets for the Treatment of Endometriosis in Adolescents Over a Treatment Period of 52 Weeks
Brief Title: Visanne Study to Assess Safety in Adolescents
Acronym: VISADO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13788; 2009-017169-53 (EudraCT Number)
Record Dates: First submitted 2011-01-25; First posted 2011-01-26 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Endometriosis
Keywords: Endometriosis; DEXA; Adolescent; Safety; Efficacy; Post-menarche
MeSH Terms: conditions — Endometriosis | interventions — dienogest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dienogest (Visanne, BAY86-5258) (Experimental): Subjects received Dienogest tablet orally at a dosage of 2 mg once daily over a period of 52 weeks.
  Interventions: Drug: Dienogest (Visanne, BAY86-5258)

INTERVENTIONS:
Drug: Dienogest (Visanne, BAY86-5258) — Subjects received Dienogest tablet orally at a dosage of 2 mg once daily over a period of 52 weeks.

SUMMARY:
A clinical trial which was designed to demonstrate the safety and efficacy of Visanne (approved in endometriosis for adults) in the adolescent population.

ELIGIBILITY:
Inclusion Criteria:

* Female adolescents after menarche (12 - less than 18 years of age) at screening. For Finland: Adolescents aged 12 - 14 years old who present with clinical features of endometriosis will only be enrolled into the study if their diagnosis of endometriosis has been confirmed by laparoscopy.
* Dysmenorrhea of at least moderate intensity, with or without chronic pelvic pain, for at least 2 cycles in the previous 4 months and one of the following conditions:

  * Clinically suspected endometriosis based on the presence of pelvic pain incompletely relieved by non steroidal anti-inflammatory drugs and/or oral contraceptives
  * Any abdominal pain associated with ultrasound findings suggestive of endometriosis (abdominal, vaginal or rectal; only after additional specific consent and assent)
  * Failure of surgical treatment for endometriosis (with cyclic or chronic pelvic pain of at least 4 months duration postsurgery)
  * Threshold for endometriosis-associated pelvic pain (EAPP) score: at least 30 on a 100 units visual analog scale retrospectively evaluated at screening for the last 4 weeks

Exclusion Criteria:

* Absence of endometriosis at laparoscopy
* Previous application of hormonal agents including oral contraceptives within 2 months, progestins, danazol within 3 months, and Gonadotropin Releasing Hormone (GnRH) agonists within 6 months prior to start of treatment
* Chronic pelvic pain that might be related to genitourinary disease or to chronic or recurrent gastrointestinal disease, including irritable bowel syndrome (defined as a disease characterized by pain relieved by defecation and irregular defecation patterns lasting at least 3 months)
* Clinically established need for primary surgical treatment of endometriosis

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 111 (Actual)
Dates: Start 2011-03; Primary Completion 2013-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Relative change in bone mineral density (BMD) of the lumbar spine as assessed by dual energy X-ray absorptiometry (DEXA) | Baseline week 52
  The measurement of BMD by DEXA is the gold standard method for investigation of bone mass.

SECONDARY OUTCOMES:
Relative Percent Change From Baseline in Whole Body Bone Mineral Density (BMD) at Week 52 Assessed by Dual-Energy X-ray Absorptiometry (DEXA) | Baseline, Week 52
  The measurement of BMD by DEXA is the gold standard method for investigation of bone mass.
Change From Baseline in Spinal Lumbar Vertebrae 2 to 4 (L2-L4) Z scores at week 52 | Baseline, Week 52
  Based on the BMD values and the weight, the age-normalized percentiles (Z-scores) were determined to allow for comparison with historical control groups. "No difference" in comparison with the historical control groups was defined as a Z-score between '-0.5' and '0.5', a lower value was defined as a value below '-0.5', and a higher value above '0.5'.
Change From Baseline in Whole Body Z-scores at Week 52 | Baseline, Week 52
  Based on the BMD values and the weight, the age-normalized percentiles (Z-scores) were determined to allow for comparison with historical control groups. "No difference" in comparison with the historical control groups was defined as a Z-score between '-0.5' and '0.5', a lower value was defined as a value below '-0.5', and a higher value above '0.5'.
Percentage of Responders at Week 24 | Week 24
  Responders were defined as subjects with reduction in pain intensity from baseline of at least 30% in the Visual Analog Scale (VAS) at Week 24. VAS consisted of a 100 unit long straight line, with verbal anchors at either end, representing a continuum of pain intensity. One end of the line with 0 score as "absence of pain" while the other end of the line with 100 score as "unbearable pain". The assessment of pelvic pain on a VAS was done once every 4 weeks till the end of the treatment (Week 52).
Change From Baseline in Pelvic Pain Over 52 Weeks Using Modified Biberoglu and Behrman Severity Profile | Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
  The cardinal symptoms inlcuded in the modified Biberoglu and Behrman severity profile were pelvic pain, dysmenorrhea, and dyspareunia (the latter only in those subjects having sexual intercourse), analyzed at all visits with symptom severity scores from 0 (none) to 3 (severe). Negative value for change from baseline indicates an improvement. In the listed categories, 'N' signifies those subjects who were evaluable for this measure.
Change From Baseline in Dysmenorrhea Over 52 Weeks Using Modified Biberoglu and Behrman Severity Profile | Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
  The cardinal symptoms inlcuded in the modified Biberoglu and Behrman severity profile were pelvic pain, dysmenorrhea, and dyspareunia (the latter only in those subjects having sexual intercourse), analyzed at all visits with symptom severity scores from 0 (none) to 3 (severe). Negative value for change from baseline indicates an improvement. In the listed categories, 'N' signifies those subjects who were evaluable for this measure.
Percentage of Subjects With Pelvic Pain Over 52 Weeks Using Modified Biberoglu and Behrman Severity Profile | Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
  In order to judge therapeutic effectiveness and to compare subjects' complaints, a severity profile score of pelvic pain was assessed using a rating scale: missing; 0 = none; 1 = mild (occasional pelvic discomfort); 2 = moderate (noticeable discomfort for most of the cycle); 3 = severe (requires strong analgesics and persists during cycle when not menstruating) based on the subject's self-assessment of symptoms. In the listed categories, 'N' signifies those subjects who were evaluable for this measure.
Percentage of Subjects With Dysmenorrhea Over 52 Weeks Using Modified Biberoglu and Behrman Severity Profile | Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
  In order to judge therapeutic effectiveness and to compare subjects' complaints, a severity profile score of dysmenorrhea was assessed using a rating scale: missing; 0 = none; 1 = mild (some loss in work efficiency); 2 = moderate (in bed part of day, occasional loss of work efficiency); 3 = severe (in bed one or more days, incapacitation) based on the subject's self-assessment of symptoms. In the listed categories, 'N' signifies those subjects who were evaluable for this measure.
Percentage of Subjects With Dyspareunia Over 52 Weeks Using Modified Biberoglu and Behrman Severity Profile | Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
  In order to judge therapeutic effectiveness and to compare subjects' complaints, a severity profile score of dyspareunia was assessed using a rating scale.
Percentage of Subjects With Pelvic Tenderness Over 52 Weeks Using Modified Biberoglu and Behrman Severity Profile | Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
  In order to judge therapeutic effectiveness and to compare subjects' complaints, a severity profile score of pelvic tenderness was assessed using a rating scale: missing; 0 = none (no pain during intercourse); 1 = mild (minimal tenderness on palpation); 2 = moderate (extensive tenderness on palpation); 3 = severe (unable to palpate because of tenderness) based on the gynecological palpation by the attending physician. In the listed categories, 'N' signifies those subjects who were evaluable for this measure.
Percentage of Subjects With Induration Over 52 Weeks Using Modified Biberoglu and Behrman Severity Profile | Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
  In order to judge therapeutic effectiveness and to compare subjects' complaints, a severity profile score of induration was assessed using a rating scale: missing; 0 = none (no pain during intercourse); 1 = mild (uterus freely mobile, induration in the cul-de-sac); 2 = moderate (thickened and indurated adnexa and cul-de-sac, restricted uterine mobility); 3 = severe (nodular adnexa and cul-de-sac, uterus frequently frozen) based on the gynecological palpation by the attending physician. In the listed categories, 'N' signifies those subjects who were evaluable for this measure.
Percentage of Subjects With Clinical Global Impression (CGI) Scores - Assessed by the Investigator | Weeks 12, 24, 36, and 52
  The investigator rating scale used in this study was based on the validated CGI scale, which is widely used as a simple tool to assess the overall effect of treatments. The investigator or a sub-investigator rated the total improvement according to the following scale: Score 1 = very much improved; Score 2 =much improved; Score 3 = minimally improved; Score 4 = no change; Score 5 = minimally worse; Score 6 = much worse; Score 7 = very much worse. None of the subjects reported Score 7. In the listed categories, 'N' signifies those subjects who were evaluable for this measure.
Percentage of Subjects With Clinical Global Impression (CGI) Scores -Assessed by the Subject | Weeks 12, 24, 36, 40, and 52
  The subject rating scale used in this study was based on the validated CGI scale, which is widely used as a simple tool to assess the overall effect of treatments. The subject was asked to rate her satisfaction with the study treatment according to the following scale: Score 1 = very much satisfied; Score 2 = much satisfied; Score 3 = minimally satisfied; Score 4 = neither satisfied nor dissatisfied; Score 5 =minimally dissatisfied; Score 6 = much dissatisfied; Score 7 = very much dissatisfied. In the listed categories, 'N' signifies those subjects who were evaluable for this measure.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (29):
- Austria (6):
  - Sankt Pölten, Lower Austria
  - Graz, Styria
  - Linz, Upper Austria
  - Graz
  - Innsbruck
  - Vienna
- Czechia (4):
  - Brno
  - České Budějovice
  - Písek
  - Prague
- Finland (3):
  - Espoo
  - Helsinki
  - Turku
- France (4):
  - Angers
  - Le Kremlin-Bicêtre
  - Paris
  - Rouen
- Germany (7):
  - Erlangen, Bavaria
  - Hamburg, Hamburg
  - Oldenburg, Lower Saxony
  - Westerstede, Lower Saxony
  - Münster, North Rhine-Westphalia
  - Lübeck, Schleswig-Holstein
  - Berlin, State of Berlin
- Spain (5):
  - Benidorm, Alicante
  - Vigo, Pontevedra
  - Seville, Sevilla
  - Valencia, Valencia
  - Seville

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu